CLINICAL TRIAL: NCT01952223
Title: A Randomized Phase III, Factorial Design, of Cabazitaxel and Pelvic Radiotherapy in Patients With Localized Prostate Cancer and High-risk Features of Relapse
Brief Title: A Phase III of Cabazitaxel and Pelvic Radiotherapy in Localized Prostate Cancer and High-risk Features of Relapse
Acronym: PEACE2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU 23 - UC-0160/1202; 2012-000566-38 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Adenocarcinoma of Prostate; Progression of Prostate Cancer
Keywords: adenocarcinoma; prostate; relapse; Radiotherapy; Androgen Deprivation Therapy; Cabazitaxel
MeSH Terms: conditions — Adenocarcinoma; Recurrence | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADT + pelvic RT (Experimental): ADT for a total duration of 3 years i.e. luteinizing hormone-releasing hormone (LHRH) agonist or LHRH antagonist +/-Peripheral anti-androgen
  Pelvic RT (by IMRT or IGRT protocol):
  * Phase 1: pelvic radiotherapy (prostate, seminal vesicles, ilio-obturator, presacral lymph nodes) (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Interventions: Radiation: Pelvic radiotherapy
- ADT + Cabazitaxel + prostate RT (Experimental): ADT Cabazitaxel: 4 CT cycles
  Prostate-only RT (IMRT or IGRT):
  * Phase 1: prostate + seminal vesicle radiotherapy (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Interventions: Drug: Cabazitaxel; Radiation: prostate radiotherapy
- ADT + cabazitaxel + pelvic RT (Experimental): ADT Cabazitaxel: 4 CT cycles
  Pelvic RT (IMRT or IGRT):
  * Phase 1: pelvic radiotherapy (prostate, seminal vesicles, ilio-obturator, presacral lymph nodes) (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Interventions: Drug: Cabazitaxel; Radiation: Pelvic radiotherapy
- ADT + prostate radiotherapy (Active Comparator): ADT for a total duration of 3 years: LHRH agonist or LHRH antagonist +/- anti-androgen
  Prostate-only RT (IMRt or IGRT):
  * Phase 1: prostate + seminal vesicle radiotherapy (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Interventions: Radiation: prostate radiotherapy

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel administered at 25 mg/m² as a 1 hour intravenous infusion every 3 weeks (1 cycle = 21 days) for 4 cycles
  Other Names: jevtana
  Arms: ADT + Cabazitaxel + prostate RT; ADT + cabazitaxel + pelvic RT
Radiation: Pelvic radiotherapy — Prostate+pelvic RT (2 Gy fractions, 5 times per week):
  * Phase 1: pelvic radiotherapy (prostate, seminal vesicles, ilio-obturator, presacral lymph nodes) (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Arms: ADT + cabazitaxel + pelvic RT; ADT + pelvic RT
Radiation: prostate radiotherapy — Prostate-only RT (2 Gy fractions, 5 times per week):
  * Phase 1: prostate + seminal vesicle radiotherapy (46 or 50 Gy according to the center)
  * Phase 2: prostate-only boost (EBRT) up to 74-78 Gy
  Arms: ADT + Cabazitaxel + prostate RT; ADT + prostate radiotherapy

SUMMARY:
The objective of this study is to assess the effect of neoadjuvant cabazitaxel and pelvic radiotherapy in combination with androgen deprivation therapy (ADT)-radiotherapy on clinical progression-free survival in patients with high-risk localized prostate cancer (with a stringent selection of patients with at least 2 high-risk features), in a 2 by 2 factorial trial.

DETAILED DESCRIPTION:
Eligible patients can be randomized via the TENALEA web site process that insure centralization of the randomization.

Randomization will be performed according a 1:1:1:1 ratio. The randomization will be stratified (by minimization) according to the number of risk factors (2 vs.3), disease extent (pN- vs. pN+ vs. pNx) and the site.

The minimization will be defined with a similar weight for all 3 stratification factors and a probability of assigning the treatment that minimize the imbalance equal to 80%.

The main analysis of progression-free survival (PFS) will be event driven (> 247 events). It will likely be performed when the median follow-up is approximately 6 years, i.e. 4 years after the inclusion of the last patient (assuming an accrual of 4 years).

A long-term analysis (allowing for robust PFS and overall survival (OS) data) will also be performed when the follow-up is approximately 10 years. Its exact timing will be discussed with the steering committee and the IDMC.

An interim analysis of the primary endpoint is planned. This interim analysis will be performed at a 0.001 level (Peto) after 50% of the events i.e. 125 have occurred.

For each comparison (CT comparison and pelvic RT comparison) the two PFS curves will be compared using the adjusted logrank test (bilateral test): adjusted logrank on pelvic RT for the CT comparison and on CT for the pelvic RT comparison. A multivariate analysis using the Cox model will also be used.

An Independent Data Monitoring Committee (IDMC) composed of international experts (at least 2 physicians and 1 statistician) will be selected.

For safety purpose, the IDMC will meet after the inclusion of 20 patients (and then again after accrual of 50 patients) in the cabazitaxel and pelvic radiotherapy arm, to assess tolerance, (i.e. after the inclusion of approximately 80 and then 200 patients in the trial). Depending on the results of this feasibility phase and of any new relevant clinical results in such a population, the remaining patients (n=848) will be enrolled.

During this second phase, the IDMC will then meet every two years approximately during accrual to carefully assess accrual rate and toxicity and examine the efficacy interim analysis results in the light of the results of similar trials.

ELIGIBILITY:
Inclusion Criteria:

1. Any T histologically confirmed adenocarcinoma of the prostate
2. No clinically or radiologically suspected metastases, including no enlarged pelvic lymph nodes (> 1 cm in small diameter)
3. Gleason score ≥ 6
4. Meets at least 2 of the following criteria for high-risk:

   * Gleason score ≥ 8
   * T3 or T4 disease (T3 defined by MRI is acceptable)
   * Prostate-specific antigen equal or greater than 20 ng/mL
5. No prior treatment for prostate cancer except lymph node dissection (patients with pN- and pN+ disease can be accrued) or ADT (started up to 6 weeks before randomization).
6. 18 years ≤ Age ≤ 75 years
7. Eastern Cooperative Oncology Group (ECOG) 0-1 performance status
8. Expected life expectancy of more than 10 years
9. Absolute neutrophil count ≥ 1.5 x 10⁹/L
10. Platelets ≥ 100 x 10⁹/L
11. Hb ≥ 9.0 g/dL
12. Hepatic function: serum bilirubin ≤ 1 upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
13. Renal function (creatinine clearance using the Chronic Kidney Disease Epidemiology group (CKD-EPI) formula ≥ 60 mL/min).
14. Potentially reproductive patients must agree to use an effective contraceptive method while on treatment and for 6 months after the final dose of investigational product.
15. Patients must be affiliated to a Social Security System or should fulfill the country legislation for clinical trials.
16. Patients who have received the information sheet and signed the informed consent form.
17. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

1. Patients with other known concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as:

   1. infection,
   2. cardiac disease such as uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within one year, left ventricular ejection fraction (LVEF) > grade 2,
   3. uncontrolled diabetes mellitus,
   4. current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, stable chronic liver disease per investigator assessment),
   5. renal disease,
   6. active GI tract ulceration, malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with active, uncontrolled ulcerative colitis are also excluded,
   7. known severely impaired lung function (spirometry and diffusing capacity of the lungs for carbon monoxide (DLCO) 70% or less of normal and O2 saturation of 88% or less at rest on room air).
2. Other prior malignancy within the last 5 years, except basal cell skin cancer
3. Physical or psychological condition that would preclude study compliance
4. Hypersensitivity to cabazitaxel (hypersensitivity reaction ≥grade 3), to other taxanes, or to any excipients of the formulation including polysorbate 80
5. Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
6. Patients who received any other investigational drugs within the 30 days prior to the start of cabazitaxel.
7. Previous pelvic irradiation that make prostatic irradiation impossible
8. Severe GI disorders precluding pelvic irradiation
9. Patients already included in another therapeutic trial involving an experimental drug
10. Individual deprived of liberty or placed under the authority of a tutor.
11. Concomitant prohibited treatment. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (see Appendix 6). A one week wash-out period is necessary for patients who are already on these treatments

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2041-07 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 10 years

SECONDARY OUTCOMES:
prostate-specific antigen response at 3 months | 10 years
biochemical progression-free survival | 10 years
metastases-free survival | 10 years
local relapse-free survival | 10 years
overall survival | 10 years
prostate cancer-specific survival | 10 years
acute toxicity | 10 years
impact of treatment on serum testosterone | 10 years
long-term toxicity | 10 years
predictive biomarkers of treatment efficacy | 10 years
quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle BOMPAS, Doctor, Principal Investigator — ICO-René Gauducheau - St Herblain; Jean-Christophe EYMARD, Doctor, Principal Investigator — Institut Jean Godinot - Reims; Guilhem ROUBAUD, Doctor, Principal Investigator — Institut Bergonié Bordeaux; Philippe BEUZEBOC, Doctor, Principal Investigator — Institut Curie Paris; Aline GUILLOT, Doctor, Principal Investigator — Institut de Cancérologie Lucien Neuwirth -ST Priest en Jarez; Claude EL KOURI, Doctor, Principal Investigator — Centre Catherine de Sienne - Nantes; Frank PRIOU, Doctor, Principal Investigator — CHD VENDEE - La Roche sur Yon; Aude FLECHON, Doctor, Principal Investigator — CENTRE LEON BERARD - lyon; Igor LATORZEFF, Doctor, Principal Investigator — Clinique Pasteur Toulouse; Karim FIZAZI, Professor, Principal Investigator — Gustave Roussy, Cancer Campus Grand Paris-Paris; Jean BERDAH, Doctor, Principal Investigator — Clinique Ste Marguerite - Hyères; Stéphane CULINE, Professor, Principal Investigator — Hôpital St Louis - Paris; Sophie ABADIE-LACOURTOISIE, Doctor, Principal Investigator — ICO - Paul Papin - Angers; Philippe FOURNERET, Doctor, Principal Investigator — Centre hospitalier de Chambéry - Chambéry; Alain GRANDGIRARD, Doctor, Principal Investigator — Centre hospitalier de Mulhouse - mulhouse; Dominique BESSON, Doctor, Principal Investigator — Clinique Armoricaine de Radiologie - St Brieuc; Loïc MOUREY, Doctor, Principal Investigator — Institut Claudius REGAUD - Toulouse; Alain RUFFION, Professor, Principal Investigator — Centre hospitalier Lyon Sud - Pierre Bénite; Tristan MAURINA, Doctor, Principal Investigator — CHRU Jean Minoz - Besançon; Pierre CLAVERE, Professor, Principal Investigator — CHU Limoges - Limoges; Véronique BECKENDORF, Doctor, Principal Investigator — Institut de Cancérologie de Lorraine; Joan Carles, Doctor, Principal Investigator — Hospital Vall d'Hebron - Barcelone; Riccardo Valdagni, Professor, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei tumori - Milan; Philippe RONCHIN, Docteur, Principal Investigator — Centre Azuréen de Cancérologie - Mougins; Eric LECHEVALLIER, Professor, Principal Investigator — Hôpital de la conception - Marseille; Gwenaëlle GRAVIS, Doctor, Principal Investigator — Institut Paoli Calmettes, Marseille; Elise CHAMPEAUX-ORANGE, Doctor, Principal Investigator — CHR Orléans La Source - Orléans; Xavier ARTIGNAN, Doctor, Principal Investigator — Saint-Gregoire Private Hospital Center; Anne DONEUX, Doctor, Principal Investigator — Clinique Générale d'Annecy; Thibaud HAASER, Doctor, Principal Investigator — Hôpital Haut L'Evèque - Pessac; Youssef TAZI, Doctor, Principal Investigator — STRASBOURG ONCOLOGIE LIBERALE - CLINIQUE SAINTE ANNE - Strasbourg; Stéphane OUDARD, Professor, Principal Investigator — HOPITAL EUROPEEN GEORGES POMPIDOU - Paris; Brigitte LAGUERRE, Doctor, Principal Investigator — CENTRE EUGENE MARQUIS - Rennes; Hakim MAHAMMEDI, Doctor, Principal Investigator — CENTRE JEAN PERRIN - Clermont Ferrand; Nadine HOUEDE, Doctor, Principal Investigator — CHRU de Nîmes Caremeau - Nîmes; Gaël DEPLANQUE, Doctor, Principal Investigator — CH Paris Saint Joseph - Paris; Marjorie BACIUCHKA-PALMARO, Doctor, Principal Investigator — Hôpital Nord Marseille; yazid BELKACEMI, Doctor, Principal Investigator — Hôpital Henri Mondor - Créteil; Mostefa BENNAMOUN, Doctor, Principal Investigator — L'Institut Mutualiste Montsouris-Paris; ali HASBINI, Doctor, Principal Investigator — Clinique Pasteur - Brest; Emmanuel GROSS, Doctor, Principal Investigator — Hôpital privé Clairval - Marseille; Bérengère NARCISO RAHARIMANANA, Doctor, Principal Investigator — CHU de TOURS Hôpital Bretonneau; Carole HELISSEY, Doctor, Principal Investigator — Hôpital d'instruction des armées Bégin - St mandé; Marta GUIX, Doctor, Principal Investigator — Hospital del Mar; Begoña PEREZ-VALDERRAMA, Doctor, Principal Investigator — Hospital Universitario Virgen del Rocio -Sevilla; Enrique GALLARDO, Doctor, Principal Investigator — Parc Tauli Sabadell Hospital Universitari - Sabadell; Maria SAEZ, Doctor, Principal Investigator — H. Virgen de la Victoria - Malaga; Montserrat DOMENECH, Doctor, Principal Investigator — Althaia, Xarxa Universitaria i assistencial de Manresa; Sergio VAZQUEZ ESTEVEZ, Doctor, Principal Investigator — H. Lucus Augusti - Lugo; Luis Miguel Anton APARICIO, Doctor, Principal Investigator — H. Teresa Herrera - Coruna; Maria José MENDEZ VIDAL, Doctor, Principal Investigator — H. Reina Sofia; Pilar LOPEZ CRIADO, Doctor, Principal Investigator — M.D. Anderson Cancer Center; Begoña MELLADO GONZALEZ, Doctor, Principal Investigator — Hospital Clinic of Barcelona; Francisco GOMEZ VEIGA, Doctor, Principal Investigator — University of Salamanca; Salvador VILLA i FREIXA, Doctor, Principal Investigator — ICO Badalona - H.U. Germans Trias; Daniel CASTELLANO, Doctor, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Institut Gustave Roussy, Villejuif, France